CLINICAL TRIAL: NCT07051031
Title: Reactogenicity, Patient Reported Outcomes and Vaccine Preference in Adults Immunized With Recombinant Protein or mRNA COVID-19 Vaccines
Brief Title: COVID-19 Reactogenicity
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Marcel Curlin (Other)
Responsible Party: Sponsor-Investigator, Marcel Curlin, Medical Director, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VBA 501
Record Dates: First submitted 2025-07-01; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Compare Post Vaccination Reactions
Keywords: COVID-19; Novavax; COVID-19 Reactogenicity; COVID-19 vaccine side effects; Novavax vs mRNA booster; Protein-based COVID vaccine; Seasonal COVID-19 booster comparison; COVID-Vaccine tolerability study; COVID-19 Post-vaccination symptoms; COVID-19 immunization study; COVID-19 Vaccine safety and daily functioning; COVID-19 Patient-reported outcomes; Novavax booster trial
MeSH Terms: conditions — COVID-19 | interventions — NVX-CoV2373 adjuvated lipid nanoparticle; BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Novavax Vaccine (Experimental): Protein-based vaccine
  Interventions: Drug: Nuvaxovid (NVX-CoV2705)
- Pfizer Vaccine (Experimental): mRNA-based vaccine
  Interventions: Drug: Pfizer-BioNTech COVID-19 vaccine

INTERVENTIONS:
Drug: Nuvaxovid (NVX-CoV2705) — COVID-19 vaccination
  Arms: Novavax Vaccine
Drug: Pfizer-BioNTech COVID-19 vaccine — COVID-19 vaccination
  Arms: Pfizer Vaccine

SUMMARY:
The purpose of this study is to compare post-vaccination reactions between the protein-based Novavax vaccine and the mRNA Pfizer vaccine. Specifically, the study aims to determine the rate of participant-reported symptoms associated with each type of vaccine.

DETAILED DESCRIPTION:
Why are we doing this study? Many people get a flu shot each year, but not as many get the COVID-19 booster, even though COVID-19 can be more serious. One reason might be that some people are worried about side effects from the vaccine.

We want to learn whether a different kind of COVID-19 vaccine, called Novavax, causes fewer side effects than the more commonly used mRNA vaccines (like Pfizer or Moderna) when given as a seasonal booster.

What is Novavax? Novavax is a protein-based COVID-19 vaccine that has been approved by the FDA. Earlier studies suggest that people may have fewer side effects with Novavax, but not many studies have directly compared it to mRNA vaccines

What is the purpose of this study? We are inviting you to join this study because you are eligible to receive a COVID-19 booster. If you choose to participate, you will receive either the Novavax vaccine or an mRNA vaccine. After your shot, we'll ask you how you feel. This helps us learn which vaccine may be easier on the body.

Why does this matter? By comparing experiences from different people, we hope to find ways to make COVID-19 boosters more acceptable and accessible. This could help more people feel confident about getting vaccinated and staying protected.

ELIGIBILITY:
Inclusion Criteria:

Adults eligible for seasonal COVID-19 vaccine, ages 18 and older Signed informed consent form (ICF) and agree to participate in the study Prior receipt of one or more COVID-19 vaccines

Exclusion Criteria:

* If a person is experiencing a moderate or severe illness or infection (as judged by the study investigator) or has a fever (temperature of 38.0°C or higher) on the day they are supposed to participate in the study, they should not join until they are feeling better and the fever is gone.
* Anyone with a medical or mental health issue, or problems with substance use that might make taking part in the study risky
* People who have had a severe allergic reaction to COVID-19 vaccines in the past
* Those who have been diagnosed with inflammation in or around the heart after receiving a COVID-19 vaccine
* Individuals who have received any other vaccine within a week before joining the study or who plan to get a vaccine on the same day as the study or within 7 days afterward

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Reactogenicity | within 7 days post vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Sciences University, Portland, Oregon, United States